CLINICAL TRIAL: NCT02907229
Title: Safety and Efficacy of Honeycomb Microporous Covered Stents (NCVC-CS1) for the Treatment of Intracranial Aneurysms: a Multicenter, Uncontrolled, Exploratory Trial
Brief Title: Safety and Efficacy of Honeycomb Microporous Covered Stents (NCVC-CS1) for the Treatment of Intracranial Aneurysms
Acronym: NCVC-CS1_UAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Kobe City General Hospital (Other); Juntendo University (Other); Kyoto University (Other)
Responsible Party: Principal Investigator, Tetsu Satow, Senior staff, National Cerebral and Cardiovascular Center, Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCVC-CS1_UAN
Record Dates: First submitted 2016-09-01; First posted 2016-09-20 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental): neuroendovascular therapy(NCVC-CS1)
  Interventions: Device: NCVC-CS1

INTERVENTIONS:
Device: NCVC-CS1 — Intervention Description

SUMMARY:
This trial is conducted to evaluate the safety and technical effectiveness of using NCVC-CS1, a newly developed honeycomb microporous covered stent, for the treatment of intracranial aneurysms which are difficult to be cured by conventional surgical or endovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

(Provisional registration)

1. Age between 20 and 75 years.
2. Target lesion is an unruptured aneurysm regardless of prior treatment diagnosed by angiography, CTA, or MRA within 180 days

   * Target aneurysm located in petrous/cavernous portion of internal carotid artery, intradural vertebral artery except for its union, or basilar artery below the orifice of superior cerebellar artery.
   * Target aneurysm is considered difficult to treat by conventional surgical/endovascular procedures
   * Target aneurysm with a sac diameter exceeding 7 mm.
   * Target aneurysm with a neck diameter over 4 mm or with a ratio "dome/neck" smaller than 2.
3. Modified Rankin score of 3 or less
4. Agreement for participating in the study and informed consent signed by the patient.

(definitive registration)

1. Target lesion must be reconfirmed by angiography or interventional procedure and is compatible with the conditions as follows:

* Target aneurysm located in petrous/cavernous portion of internal carotid artery, intradural vertebral artery except for its union, or basilar artery below the orifice of superior cerebellar artery.
* Target aneurysm is considered difficult to treat by conventional surgical/endovascular procedures
* Target aneurysm with a sac diameter exceeding 7 mm.
* Target aneurysm with a neck diameter over 4 mm or with a ratio "dome/neck" smaller than 2.
* Parent artery of target aneurysm is accessible by the investigational devices
* The diameter of the parent artery between 3.5 and 5 mm.

Exclusion Criteria:

(Provisional registration)

1. Any invasive surgical procedure within 30 days before registration.
2. Prior stent implantation at the site of target aneurysm
3. Existence of intracranial tumor, arteriovenous malformation for which any intervention is considered necessary, or co-existence of unruptured intracranial aneurysm whose sac diameter over 5mm within the target vessel.
4. Coexistence of other unruptured intracranial aneurysms which are planned for intervention
5. Target vessel not suitable for delivery and placement of covered stent because of anatomical configuration (i.e. severe bend or tortuosity).
6. More than 50% stenosis in the target vessel or its proximity including extracranial region.
7. Any intracranial hemorrhage within 42 days before registration.
8. Co-morbid conditions that may limit survival to less than 6 months, or difficult to observe the patient for 6 months.
9. Renal dysfunction whose serum creatinine more than 2.0
10. Contraindications to antiplatelet or anticoagulant treatment because of allergy or hemorrhagic diathesis.
11. Platelets less than 100,000/mm3 or known dysfunction of platelets.
12. Active bacterial infection.
13. Any cardiac, hematological, intracranial, or vessel disease which are considered to have high risk of neurological events (severe cardiac failure, atrial fibrillation, arteritis, known carotid artery stenosis, etc.).
14. History of severe allergy to contrast dye.
15. Known allergy to cobalt-chromium alloy and polyurethane. clopidogrel, heparin, nitinol, local or general anesthesia
16. Subjects who have enrolled, or are planned to participate in other clinical trial or intervention study.
17. Pregnant woman
18. Unsuitable patients judged by the physician attending this trial.

(definitive registration)

1. History of any invasive surgical procedure after the provisional registration.
2. Any new neurological signs within 24 hours prior to the procedure.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: Any stroke or death related to the procedure within 180 days | 180 days after the procedure
Efficacy evaluation: Complete obliteration of target aneurysm and patency of target vessel (less than 50% stenosis) confirmed by angiography at 180 days after the procedure | 180 days after the procedure

SECONDARY OUTCOMES:
Technical success (stent placement in the target lesion covering aneurysmal neck without occlusion of target vessel) | 180 days after the procedure
Any death within 180 days after the procedure | 180 days after the procedure
Any death by neurological reason within 180 days after the procedure | 180 days after the procedure
Any adverse event or adverse device effect | 180 days after the procedure
Neurological assessment (scale ; mRS) | 180 days after the procedure
Neurological assessment (scale ; Barthel Index) | 180 days after the procedure
Neurological assessment (scale ; NIHSS) | 30 days after the procedure
Neurological assessment (scale ; GCS) | 30 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tetsu Satow, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (4):
- Japan (4):
  - Kobe City General Hospital, Kobe, Hyōgo
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kyoto University Hospital, Kyoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamamoto H, Hamasaki T, Onda K, Nakayama Y, Ishii A, Oishi H, Sakai N, Satow T. Evaluating the safety and technical effectiveness of a newly developed intravascular 'flow isolator' stent for the treatment of intracranial aneurysms: study protocol for a first-in-human single-arm multiple-site clinical trial in Japan. BMJ Open. 2019 May 9;9(5):e020966. doi: 10.1136/bmjopen-2017-020966. PMID 31072845